CLINICAL TRIAL: NCT01917305
Title: Influence of Platform-switching on Bone Level Alterations: a 3 Year RCT.
Brief Title: Influence of Platform-switching on Bone Level Alterations: a 3 Year Randomized Clinical Trial (RCT).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Søren Jepsen (Other)
Responsible Party: Sponsor-Investigator, Søren Jepsen, Professor Dr.med Dr. med.dent MS, Chair, University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFS3YRCT
Record Dates: First submitted 2013-07-31; First posted 2013-08-06 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Periimplant Crestal Bone Level Changes
Keywords: Bacteria; bone level; bone loss; dental implants; implant design; platform-shifting; platform-matching
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- platform-switched implant (Experimental): platform-switched implant
  Interventions: Device: platform-shifted implant
- platform-matched implant (Active Comparator): platform-matched implant
  Interventions: Device: platform-shifted implant

INTERVENTIONS:
Device: platform-shifted implant

SUMMARY:
The concept of platform-switching has been introduced to implant dentistry based on clinical observations of reduced periimplant crestal bone loss. However, published available data are controversial and most studies are limited to 12 months. The aim of the present RCT was to test the hypothesis that platform-switching has a positive impact on crestal bone level changes after 3 years.

DETAILED DESCRIPTION:
Two implants with a diameter of 4 mm were inserted crestally in the posterior mandible of 25 subjects. After three months of submerged healing, single-tooth crowns were randomly placed, either with (3.3mm platform, test) or without platform-switching (4mm platform, control). Patients were followed up at short intervals for monitoring of healing an oral hygiene. Statistical analysis for the influence of time and platform-type on bone levels employed the Brunner-Langer Model.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* edentulous gap in the posterior mandible for placement of 2 implants
* sufficient bone height above the alveolar nerve for placement of implants with a height of 9.5mm
* bone width for placement of implants with diameter of 4mm
* at least 4mm keratinized mucosa
* medium or a thick soft tissue biotype

Exclusion Criteria:

* infectious disease
* diabetes or osteopathy
* active periodontitis
* medication influencing bone metabolism
* lactating or pregnant women

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change of vertical implant bone level | Implant insertion (baseline), 3 months (reopening), 4 months (crown mounting), 12, 25 and 38 months

SECONDARY OUTCOMES:
probing depths | 4, 8, 12, 25, 38 months
Bleeding | baseline, 4, 8, 12, 25, 38 months
Plaque | baseline, 4, 8, 12, 25, 38 months

REFERENCES:
- [Derived] Jervoe-Storm PM, Hablutzel AS, Bartels P, Kraus D, Jepsen S, Enkling N. Comparison of irrigation protocols for the internal decontamination of dental implants-results of in vitro and in vivo studies. Clin Oral Implants Res. 2021 Oct;32(10):1168-1175. doi: 10.1111/clr.13814. Epub 2021 Aug 27. PMID 34352143
- [Derived] Enkling N, Johren P, Katsoulis J, Bayer S, Jervoe-Storm PM, Mericske-Stern R, Jepsen S. Influence of platform switching on bone-level alterations: a three-year randomized clinical trial. J Dent Res. 2013 Dec;92(12 Suppl):139S-45S. doi: 10.1177/0022034513504953. Epub 2013 Oct 24. PMID 24158333